CLINICAL TRIAL: NCT04218565
Title: Efficacy and Safety of Golimumab in the Treatment of Refractory Uveitis in Patients With Behcet's Disease
Brief Title: Golimumab for the Treatment of Refractory Behcet's Uveitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: only one patient enrolled
Sponsor: Wenjie Zheng (Other)
Responsible Party: Sponsor-Investigator, Wenjie Zheng, Professor， Department of Rheumatology, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOL-BDU-PUMCH
Record Dates: First submitted 2019-12-08; First posted 2020-01-06 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Behcet Syndrome; Uveitis
MeSH Terms: conditions — Behcet Syndrome; Uveitis | interventions — golimumab

STUDY DESIGN:
Intervention Model Description: Golimumab is approved for the treatment of several inflammatory diseases, the self-control study aims to evaluate the response to GOL in refractory BDU.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Golimumab for refractory BDU (Experimental): This study is a self-control study and all the participants will be enrolled in the interventional arm.
  Interventions: Biological: Golimumab (GOL)

INTERVENTIONS:
Biological: Golimumab (GOL) — Patients with refractory BD associated uveitis will receive Golimumab therapy, the efficacy and corticosteroids-sparing effects will be evaluated.

SUMMARY:
The aim of this single-center prospective study is to evaluate the efficacy and safety of Golimumab （GOL）, fully humanized anti-tumor necrosis factor (TNF)-α monoclonal antibody, in the treatment of refractory Uveitis of Behçet's disease (BDU), to verify its effects on decreasing the dose of cortical steroids, and to determine whether it can reduce BDU recurrence.

DETAILED DESCRIPTION:
Uveitis of Behçet's disease (BDU) is the most common form of ocular manifestations, which is also the leading cause of irreversible visual impairment. The aim of the study is to improve the treatment strategy of the disease as well as to reduce blindness.

Monoclonal anti-TNF antibodies were recommended in 2018 recommendations for treating eye involvement affecting the posterior segment (level of evidence: IIA; strength of recommendation: B), Infliximab was mentioned for the treatment of initial or recurrent episode of acute sight-threatening uveitis.

Golimumab （GOL）is a fully-humanized anti-TNF-α monoclonal antibody, retrospective study on non-infectious uveitis and BDU has obtained promising results.

This single-center prospective study is to evaluate the efficacy and safety of GOL in the treatment of refractory BDU, to verify its effects on tapering the dose of corticosteroids, and to determine whether it can reduce BDU recurrence. We aim to enroll nine refractory BDU patients with acute onset posterior uveitis, with difficulty tapering corticosteroids while being treated with at least one of the commonly used immunosuppressants.

All participants will receive GOL monthly for six months, oral immunosuppressants will remain unchanged. During follow-up, intraocular inflammation status, BCVA, as well as extraocular manifestations, will be recorded. The primary endpoints are the efficacy of the first dose of GOL, and the recurrence of uveitis after 12 months of treatment. Secondary endpoints other than intraocular inflammation will be achieved on each follow-up visit, as the quality of life improvements, side effects, recurrence of uveitis, and corticosteroids-tapering effects.

On statistical analysis, the self-control treatment efficiency and recurrence rate difference will be determined using T-test of paired samples at a significance level of 0.05(2-sided).

To ensure the interest of the participants, our study has been reviewed by the ethics committee, and drug clinical research liability insurance was prepared.

ELIGIBILITY:
Inclusion Criteria:

* All participants fulfill the proposed International Criteria for BD, either ISG (International Study Group) criteria(1990) or ICBD(International Conference on Behcet's Disease) criteria(2013).
* All participants present with refractory BDU, acute onset uveitis, either posterior segment involvement or panuveitis, with difficulty tapering corticosteroids while being treated with at least one of the commonly used immunosuppressants, without severe extraocular manifestations.

Exclusion Criteria:

* Patients with impaired hepatic and renal function, other severe ocular diseases, active tuberculosis, viral hepatitis, malignancy, pregnancy, congestive heart failure, or had biologics treatment within three months will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Efficacy of Golimumab on BD Uveitis | four weeks
  Efficacy of Golimumab based on Behçet's disease ocular attack score 24 （BOS24）
Efficacy of Golimumab on BD Uveitis | four weeks
  Efficacy of Golimumab based on Best corrected visual acuity(BCVA)
Efficacy of Golimumab on BD Uveitis | four weeks
  Efficacy of Golimumab based on Optical Coherence tomography(OCT)).
Difference of recurrence rate before and after intervention | 12 months
  Difference of recurrence rate of uveitis before and after 12 months of GOL treatment

SECONDARY OUTCOMES:
Intraocular inflammation evaluation BOS24 index | each follow-up visit / every four weeks, up to six months
  Visual acuity, anterior chamber cells, vitreous opacities, retinal inflammation, macular thickness, etc.
Corticosteroid-tapering effects | six months
  Corticosteroid will be tapered to minimum dose(Prednisone 5-10mg/d) within four months during the course of GOL treatment.
Changes of uveitis recurrence | six months
  Changes of recurrence rate before and after six months of GOL treatment.
Severity of uveitis on recurrence | six months
  Differences of severity of recurrence before and after treatment, measured by BOS24.
Severity of uveitis on recurrence | six months
  Differences of severity of recurrence before and after treatment, measured by , BCVA.
Severity of uveitis on recurrence | six months
  Differences of severity of recurrence before and after treatment, measured by OCT.
Impact on quality of life | each follow-up visit / every four weeks, up to six months
  Record quality of life on questionnaire, BehÇet's disease current activity form 2006（BDCAF2006）.
Impact on quality of life | each follow-up visit / every four weeks, up to six months
  Record quality of life on questionnaire, short from Health Survey(SF-36).
Side effects of treatment | six months
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Wenjie Zheng, M.D., Principal Investigator — Department of Rheumatology, Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No